CLINICAL TRIAL: NCT03298282
Title: Integrated Coronary Multicenter Imaging Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2017-0049
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imaging Registry: Imaging cohort: Patients with intermediate lesions
  Interventions: Other: OCT (Optical Coherence Tomography); Other: Coronary CTA; Other: FFR

INTERVENTIONS:
Other: OCT (Optical Coherence Tomography) — Coronary images by OCT and selective CTA and FFR values will be registered.
Other: Coronary CTA — Coronary images by OCT and Coronary CTA and FFR values will be registered.
Other: FFR — Coronary images by OCT and selective CTA and FFR values will be registered.

SUMMARY:
The coronary images of selective angiography and optical coherence tomography with FFR(Fractional Flow Reserve) values of the intermediate lesions (40-70% stenosis) will be prospectively registered.

DETAILED DESCRIPTION:
The patients with intermediate lesions after CT angiography and invasive coronary angiography will be screened, and optical coherence tomography, FFR and selective CT angiography will be performed. The coronary images and FFR values will be registered, and the patients will be followed-up up to 2 years to investigate the adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent coronary CT angiography because of chest pain
* Patients who need OCT or FFR evaluation because of intermediate lesions according to invasive angiography (diameter stenosis of 40-70%)
* Age: 20-80 yrs
* Patients who consent and fully understand the protocol
* Patients who consent the clinical follow-up
* Patients who can be followed-up

Exclusion Criteria:

* Patients who had contrast allergy
* Patients who had unstable blood pressure needing the vasopressors
* Patients who had severe left ventricular function (left ventricular ejection fraction<30%)
* Chronic kidney disease who had Cr level of greater than 2.0 mg/dl
* Patients whose expected survival is less than 12 months
* Patients who had a severe valvular disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary cardiovascular hospital
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of plaque on coronary CTA for during 2 years | at registration
Change of plaque on coronary CTA for during 2 years | at 2-year follow up
Change of plaque on coronary OCT for during 2 years | at registration
Change of plaque on coronary OCT for during 2 years | at 2-year follow up
Change of FFR value during 2 years | at registration
Change of FFR value during 2 years | at 2-year follow up
Comparison of computational FFR derived from OCT to invasive FFR | at registration
Comparison of computational FFR derived from OCT to invasive FFR | at 2-year follow up

SECONDARY OUTCOMES:
Adverse event for 2 years (myocardial infarction, cardiovascular death) | within 2 years after registration
Power of plaque characteristics on coronary CTA for predicting adverse events | within 2 years after registration
Power of plaque characteristics on OCT for predicting adverse events | within 2 years after registration

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Cardiovascular Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YJ, Kim YW, Ha J, Kim M, Guagliumi G, Granada JF, Lee SG, Lee JJ, Cho YK, Yoon HJ, Lee JH, Kim U, Jang JY, Oh SJ, Lee SJ, Hong SJ, Ahn CM, Kim BK, Chang HJ, Ko YG, Choi D, Hong MK, Jang Y, Lee JS, Kim JS. Computational Fractional Flow Reserve From Coronary Computed Tomography Angiography-Optical Coherence Tomography Fusion Images in Assessing Functionally Significant Coronary Stenosis. Front Cardiovasc Med. 2022 Jun 13;9:925414. doi: 10.3389/fcvm.2022.925414. eCollection 2022. PMID 35770218